CLINICAL TRIAL: NCT04016467
Title: The Effect of Thoracic Spinal Manipulation on Vulvar Vestibule Pain: a Controlled Clinical Study
Brief Title: Effect of Spinal Manipulation on Vulvar Pain
Acronym: SpManipPP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of participants in available recruitment area
Sponsor: University of Mary Hardin-Baylor (Other)
Collaborators: Integrity Rehab and Home Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 6.7.2018
Record Dates: First submitted 2019-07-01; First posted 2019-07-11 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Vulvodynia; Perineal Pain; Vulvar Pain
Keywords: Spinal Manipulation
MeSH Terms: conditions — Vulvodynia

STUDY DESIGN:
Intervention Model Description: Controlled clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomized intervention, blinding of pain measure to intervention PT, and blinding of intervention assignment pain assessment PT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracic Manipulation (ThM) (Experimental): Will undergo spinal manipulation between pain assessment pre and post.
  Interventions: Other: Thoracic manipulation
- Sham thoracic treatment (ThS) (Sham Comparator): Sham manipulation between pain assessment pre and post
  Interventions: Other: Sham thoracic treatment

INTERVENTIONS:
Other: Thoracic manipulation — High velocity, small amplitude thrust treatment to spine that elicits a neurophysiologic response.
  Arms: Thoracic Manipulation (ThM)
Other: Sham thoracic treatment — Hand placement on thorax without thrust.
  Arms: Sham thoracic treatment (ThS)

SUMMARY:
The purpose of the study is to determine the effect of thoracic spine manipulation on vestibule pain as determined by sensory testing (q-tip and pressure algometry) in a group of women with provoked vestibulodynia (PVD). The objective is to compare the immediate effect of manipulation and sham manipulation on the results of sensory testing of the external vulva, or vestibule.

DETAILED DESCRIPTION:
PRE-SCREENING: Participants expressing interest in this study will be interviewed to determine if eligibility criteria to participate in this study are met. If that is the case, the participant will then be invited to attend the familiarization and study session and informed of the need to refrain from alcohol use and keep medication regiment consistent in the 24 hours prior to the study appointment.

FAMILIARIZATION and CONSENT: During this session, the study protocol will be described and a written explanation of the study provided to the participant. After any questions have been addressed, the participant will sign the informed consent statement. Next, the participant will complete demographic and health questionnaires, which will be reviewed by the investigators to ensure eligibility criteria are met. If qualified,the participant will complete additional questionnaires that ask about pain, other symptoms of the pelvis and perineum and about feelings of anxiety and depression. Along with the questionnaires, a pelvic and lower extremity secondary screening examination will be performed as described below.

SECONDARY SCREEN and BASELINE TESTING: During the lower extremity screening examination, the participant will be asked to bend and straighten their spine, stretch in specific ways with the spine and legs and report if these motions provoked discomfort or pain. The pelvic exam and baseline testing is to ensure that the participant has pain in the perineum (area that is wiped after toileting). This will be tested in 2 ways, one using a sterile cotton tipped swab (q-tip test) and the other with a pressure sensing device called an algometer. One trained pelvic floor Physical Therapist (PT1) investigator will perform these tests. While investigator PT1 waits outside, the participant will undress from the waist down then lay under a sheet. PT1 will enter and perform the sensory tests during which the participant's pelvic floor and vestibule will be exposed in a similar manner to receiving a gynecologic exam. PT1 will use a q-tip to touch specific points around the vaginal opening (vestibule) and ask the participant to report any pain on a scale of 0 (none)-10 (worst). Next, a pressure algometer will be used to measure the amount of pressure tolerated on the most painful q-tip spot. This algometer has a flat disc, the size of a pencil eraser, that is covered to ensure cleanliness. Then the participant's lower body will be draped. Participant's with provoked pain are eligible to continue; those without are not eligible to continue in the study and will be done.

INTERVENTION and REPEAT BASELINE TESTING: The eligible participants are randomly assigned, by participant number, into one of the two testing groups. One group will receive a sham thoracic spine manipulation (ThS) and the other, a thoracic spine manipulation (ThM). During the thoracic intervention, the participant will lay on their back with arms crossed. The second PT (PT2), who is blinded to the results of the pain testing, will position one hand along the participant's thoracic spine and the other on the participant's crossed arms to apply a posterior motion to the participant's spine. This will be small motion that may be done quickly or slowly. After the technique, the participant will continue to rest on their back, while PT1 returns to repeat testing of the vestibule with the q-tip and algometer in the same manner as previously described. Then participation is finished.

ELIGIBILITY:
Inclusion Criteria:

* Provides written and dated informed consent to participate in the study.
* Is between the ages of 18-40 years.
* Reports pain in the pelvis and/or vestibule (area that is wiped after using the toilet) that has been present for ≥ 6 weeks.
* Has not had treatment for pelvic or vestibule pain in the 6 months prior to study participation.
* Is willing and able to comply with study protocol.
* Is healthy and free from disease, as determined by a health history questionnaire and screening exam.
* Agrees to abstain from alcohol consumption 24 hours prior to the study protocol.
* Reports a consistent regimen of pain medication use in the 6 weeks prior to the study protocol. This includes both prescription and over the counter medications.
* Secondary Inclusion Criteria: demonstrates provoked vestibule pain to q-tip testing.

Exclusion Criteria:

* Is currently pregnant, or attempting to become pregnant, as the intervention is contraindicated for this population.
* Fails the health history, spine screen; or does not demonstrate provoked vestibule pain with q-tip test.
* Has undergone any spine or pelvic girdle surgery in the 12 months prior to the study.
* Has ever had sling/mesh placement to the pelvic region.
* Has been diagnosed with osteopenia, osteoporosis, acute infection or arthritis flare, or other condition that could weaken the bony skeleton.
* Has ever had a thoracic spine fracture.
* Has had a change in any prescription or over-the-counter medications used for pain in the 6 weeks prior to the study.
* Any other condition or adverse event in which study investigator recommend removal from the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Change in Numeric Pain Rating Scale (NPRS) (0=none to 10=worst) report to cotton swab test in clock pattern | Pre and immediately post thoracic intervention. No longer term follow-up is planned.
  Participant report on NPRS

SECONDARY OUTCOMES:
Change in peak pressure algometer | Pre and immediately post thoracic intervention. No longer term follow-up is planned
  Nm2 pressure reading of provoked pain on most painful point

CONTACTS AND LOCATIONS:
Overall Officials: PATRICIA NELSON, PT, ScD, Principal Investigator — University of Mary Hardin-Baylor
Locations (1):
- Integrity Rehab and Home Health, Copperas Cove, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No data sharing is planned